CLINICAL TRIAL: NCT02578719
Title: Placebo-Controlled Randomized Double Blind Trial of Blocking Greater Occipital Nerve Block With Bupivacaine Versus Saline in the Treatment of Chronic Migraine
Brief Title: Greater Occipital Nerve (GON) Block Effectivity in the Treatment of Chronic Migraine: 6 Months Follow up
Acronym: GON
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Local Drug Authority didn't give permission to start.
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Levent E. Inan, Professor, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B.10.4.ISM.4.06.68.49/
Record Dates: First submitted 2015-10-08; First posted 2015-10-19 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- drug: bupivacaine (Placebo Comparator): Placebo comparator: bupivacaine first 3 months 0.5% 1 cc bupivacaine diluated with 1.5 cc saline enjection will be used in GON block once a month. If effectiveness is proved then blindness will be opened and all patients will be blocked by 0.5% 1 cc bupivacaine diluated with 1.5 cc saline once a month for 3 months.
  Interventions: Drug: bupivacaine
- placebo (Placebo Comparator): first 3 months 2.5 cc saline enjection will be used in GON block once a month. If effectiveness is proved then blindness will be opened and all patients will be blocked by 0.5% 1 cc bupivacaine diluated with 1.5 cc saline once a month for 3 months.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: bupivacaine — marcaine %0.5 20 ml flacon
  Other Names: marcaine
  Arms: drug: bupivacaine
Drug: saline — %0.9 sodium chloride
  Other Names: %0.9 sodium chloride
  Arms: placebo

SUMMARY:
This study evaluates effectiveness of greater occipital nerve blocks with bupivacaine compared to placebo in chronic migraine patients.

DETAILED DESCRIPTION:
The greater occipital nerve (GON), which derives most of its fibers from the C2 dorsal root, is the primary sensory nerve of the occipital region. The response to GON blockade was not simply dependent on the direct local anesthetic effect of the injection . The mechanism of action might have been via changes in brain nociceptive pathways. Another possible explanation for these findings is, therefore, that GON injections initiated diffuse noxious inhibitory controls, independent of anesthetic effect . Neurophysiological and clinical data suggest there is a functional connection between the sensory occipital segments and the trigeminal nociceptive system in humans.

ELIGIBILITY:
Inclusion Criteria:

* Chronic migraine headache according to International Headache Society Classification Criteria
* Patients who are not using any prophylacting agent

Exclusion Criteria:

* patients given similar treatments before
* pregnant women
* hereditary diseases causing bleeding
* patients who have intracranial tumor or operation in posterior fossa
* allergic reactions to local anesthetics.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
50% decrease in migraine severity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Levent E Inan, Prof., Principal Investigator — Bozok University Neurology Department

REFERENCES:
- [Background] Inan LE, Inan N, Karadas O, Gul HL, Erdemoglu AK, Turkel Y, Akyol A. Greater occipital nerve blockade for the treatment of chronic migraine: a randomized, multicenter, double-blind, and placebo-controlled study. Acta Neurol Scand. 2015 Oct;132(4):270-7. doi: 10.1111/ane.12393. Epub 2015 Mar 13. PMID 25765043